CLINICAL TRIAL: NCT00134732
Title: Assess the Immunogenicity, Safety & Reactogenicity of 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants (6-12 Weeks of Age at First Dose) Previously Uninfected With Human Rotavirus
Brief Title: Study of 2 Doses of Oral Live Attenuated Human Rotavirus (HRV) Vaccine for the Prophylaxis of Rotavirus Gastroenteritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 103478
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
Keywords: Prophylaxis of Rotavirus Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: Live attenuated human rotavirus vaccine

SUMMARY:
Rotavirus (RV) is the most important cause of acute gastroenteritis (GE) requiring the hospitalization of infants and young children in developed and developing countries and can be a frequent cause of death in children less than 5 years of age (estimated nearly 500,000 annual deaths worldwide). GlaxoSmithKline (GSK) Biologicals has developed a vaccine against human rotavirus gastroenteritis. This study will provide data for Korean regulatory authorities about the immunogenicity and safety of this vaccine in Korean children aged 2 months at the time of the first dose.

DETAILED DESCRIPTION:
The study consists of two groups of children recruited in different centers in Korea. One group will receive the HRV vaccine and one group will receive the placebo. The vaccine or placebo will be administered starting at 2 months of age according to a two dose schedule (0, 2 months). The study will consist of three visits. At the first visit, one blood sample will be taken before vaccination and the first dose will be administered. At the second visit (2 months after first dose), the second vaccine will be administered. At the third visit (2 months after second dose), a blood sample will be taken. A 15-day (Day 0 - 14) follow-up period will be observed for general symptoms solicited in the study (fever, fussiness/irritability, diarrhea, vomiting, loss of appetite and cough/runny nose). A 43-day (Day 0 - 42) follow-up will be observed for other unsolicited symptoms. Serious adverse events will be followed-up throughout the study. A stool sample should be collected from the child at any point during the study if he/she develops any GE.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems, as established by medical history and physical examination, before entering into the study.
* Subjects for whom the vaccination history is available from vaccination diary cards or medical charts or patient diary cards.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine or placebo, or planned use during the study period.
* Planned administration of a vaccine (including routine paediatric vaccines) not foreseen by the study protocol during the period starting from 14 days before each dose of study vaccine(s) and ending 14 days after.
* Any clinically significant history of chronic gastrointestinal (GI) disease including any uncorrected congenital malformation of the GI tract or other serious medical condition, as determined by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required).
* Major congenital defects or serious chronic illnesses such as malignant disease (e.g. melanotic neuroectodermal tumor, malignant rhabdoid tumor, etc.), serious atopic dermatitis, conditions that are the result of premature birth, etc.
* Acute disease at time of enrolment. (Acute disease is defined as the presence of moderate or severe illness with or without fever i.e. temperature >= 37.5°C as measured by an axillary thermometer or >= 38.0°C as measured by a rectal thermometer. A temperature greater than or equal to these cut-offs warrants deferral of the vaccination pending recovery of the subject.)
* GE within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period. Oral intake of immunoglobulins via, e.g., breastfeeding is allowed.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth. (For corticosteroids, this will mean prednisone, or equivalent, >= 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Previous confirmed occurrence of RV GE.
* Household contact with an immunosuppressed individual

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150
Dates: Start 2005-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Percent who seroconverted (anti-rota serum IgA, 2 months post dose 2)

SECONDARY OUTCOMES:
Grade 2 and 3 fever, vomiting, diarrhea, solicited symptoms
Unsolicited events
Serious adverse events (SAEs)
Presence of rota in GE tools
Concentration IgA 2 months post dose 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- South Korea (4):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 103478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register